CLINICAL TRIAL: NCT00302965
Title: Effectiveness of Fresh Frozen Plasma in Critical Care (EPICC) Trial
Brief Title: Effectiveness of Plasma Transfusions in Critical Care Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2004341-01
Record Dates: First submitted 2005-09-13; First posted 2006-03-15 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Coagulation
Keywords: Plasma; Trauma; Critical Care
MeSH Terms: conditions — Thrombosis; Wounds and Injuries

INTERVENTIONS:
Drug: Frozen Plasma

SUMMARY:
Measuring the effectiveness of plasma transfusions in critical care

DETAILED DESCRIPTION:
Measuring the effectiveness of plasma transfusions in critical care

ELIGIBILITY:
Inclusion Criteria:

* ICU Admission
* INR > 1.2
* Require FFP for active bleeding and/or prior to an invasive procedure
* Are able to provide consent or proxy consent

Exclusion Criteria:

* Congenital or acquired coagulation factor deficiency
* Platelet count < 50 x 109 /L and have NOT received subsequent platelet transfusion
* Consumptive coagulopathy (bleeding ≥ 3 sites and ↓ plts, ↓ fib, ↑ d dimer)
* Uncontrolled bleeding (6 or more units of blood in the last 6 hours)
* Receiving therapeutic doses of heparin/heparinoid (must be off for at least 6 hours)
* Have received clotting factor concentrates in the previous 24 hours
* Are expected to require surgery in the next 48 hours
* Survival expected to be less than 48 hours
* Currently enrolled in another study with a similar outcome
* Previous enrollment in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with a correction of the INR (Determined by the treating physician)
Secondary outcomes include changes in coagulation tests (INR, aPTT and individual coagulation factor levels
bleeding and complications from FFP (fluid overload, transfusion reactions).

SECONDARY OUTCOMES:
Secondary outcomes include changes in coagulation tests (INR, aPTT and individual coagulation factor levels
bleeding and complications from FFP (fluid overload, transfusion reactions).

CONTACTS AND LOCATIONS:
Overall Officials: Alan Tinmouth, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada